CLINICAL TRIAL: NCT00147758
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of WelChol® in Type 2 Diabetics With Inadequate Glycemic Control on Sulfonylurea Monotherapy or Sulfonylurea Therapy in Combination With Other Oral Anti-Diabetic Agents
Brief Title: WelChol® and Sulfonylurea in Treating Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-303
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Colesevelam Hydrochloride

INTERVENTIONS:
Drug: Colesevelam hydrochloride

SUMMARY:
The purpose of the study is to see how safe and effective and tolerable the use of colesevelam hydrochloride is for type 2 diabetes when added to sulfonylurea alone or in combination with other anti-diabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, inclusive
* Diagnosed with type 2 diabetes
* Stable dose of sulfonylurea alone or in combination with other anti-diabetic medications for 90 days
* Hemoglobin A1c value 7.5% to 9.5%, inclusive
* C peptide > 0.5 ng/mL
* Prescribed ADA diet

Exclusion Criteria:

* History of type 1 diabetes or ketoacidosis
* History of pancreatitis
* Uncontrolled hypertension
* Allergy or toxic response to colesevelam or any of its components
* Serum LDL-C < 60 mg/dL
* Serum TG > 500 mg/dL
* Body mass index (BMI) > 45 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To assess the additional lowering of HbA1c achieved by addition of colesevelam hydrochloride to current antidiabetic therapy

SECONDARY OUTCOMES:
To assess the fasting plasma glucose and fructosamine lowering efficacy;
To assess glycemic control response rate;
To assess the improvement in insulin sensitivity;
To assess the effect on C reactive protein;
To assess lipids and lipoproteins;
To assess the safety and tolerability of colesevelam hydrochloride as add-on therapy

CONTACTS AND LOCATIONS:
Locations (47):
- United States (45):
  - Birmingham, Alabama
  - Tuscumbia, Alabama
  - Little Rock, Arkansas
  - Searcy, Arkansas
  - Concord, California
  - Irvine, California
  - La Jolla, California
  - Los Angeles, California
  - Los Gatos, California
  - West Hills, California
  - Coral Gables, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Pembroke Pines, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Kansas City, Missouri
  - St Louis, Missouri
  - Rochester, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Marion, Ohio
  - Perrysburg, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Charleston, South Carolina
  - Bristol, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Arlington, Virginia
  - Richmond, Virginia
  - Lakewood, Washington
  - Renton, Washington
- Mexico City, Mexico
- Lima, Peru

REFERENCES:
- [Derived] Fonseca VA, Rosenstock J, Wang AC, Truitt KE, Jones MR. Colesevelam HCl improves glycemic control and reduces LDL cholesterol in patients with inadequately controlled type 2 diabetes on sulfonylurea-based therapy. Diabetes Care. 2008 Aug;31(8):1479-84. doi: 10.2337/dc08-0283. Epub 2008 May 5. PMID 18458145